CLINICAL TRIAL: NCT05393089
Title: A Phase 2, Multicenter, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety and Efficacy of AGN-190584 in Subjects With Pseudophakic Presbyopia
Brief Title: Study of AGN-190584 Eye Drops to Assess Safety and Efficacy in Participants Aged 40-80 Years With Pseudophakic Presbyopia
Acronym: ARIES
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M21-194
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Presbyopia
Keywords: Presbyopia; Pseudophakic Presbyopia; AGN-190584; ARIES; Pilocarpine HCl
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AGN-190584 (Experimental): Participants will receive one drop of AGN-190584 instilled in each eye once daily for 14 days.
  Interventions: Drug: AGN-190584
- Vehicle (Placebo Comparator): Participants will receive one drop of vehicle instilled in each eye once daily for 14 days.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: AGN-190584 — Eye drops
  Arms: AGN-190584
Drug: Vehicle — Eye drops
  Arms: Vehicle

SUMMARY:
Presbyopia is a condition in which the eye exhibits a diminished ability to focus on near objects with increasing age. This study will assess the safety and exploratory efficacy of AGN-190584 is in treating participants with pseudophakic presbyopia.

AGN-190584 is approved (in the United States) for use in adults with presbyopia (including those who are pseudophakic) and this study is being conducted to better understand the safety and efficacy in the pseudophakic presbyopia population. This study is double-masked meaning that neither the participants nor the study doctors will know who will be given AGN-190584 and who will be given vehicle (does not contain treatment drug). Study doctors put the participants in 1 of the 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 3 chance that participants will be assigned to vehicle. Approximately 150 participants aged 40-80 years with pseudophakic presbyopia will be enrolled in approximately 30 sites in the US.

Participants will receive eye drops of AGN-190584 or vehicle once daily in the morning in each eye for 14 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study. The effect of the treatment will be evaluated by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* History of bilateral pseudophakia with monofocal intraocular lenses corrected for distance (noncomplicated cataract surgery), with identifiable intraocular lens type/brand, at least 3 months after surgery (prior to baseline), and be in stable condition.
* If a participant has had neodymium-doped yttrium aluminum garnet (Nd:YAG) laser capsulotomy, it needs to be done bilaterally at least 1 month prior to baseline.
* Subjective complaints of poor near vision that impacts activities of daily living, as defined by at least a moderate impact (score >= 3) on at least 1 question on 25-Item National Eye Institute Visual Function Questionnaire (NEI VFQ-25) Questions 5 to 7 in the main questionnaire or Near Vision Subscale, Questions A3 to A5 in the Appendix of Optional Additional Questions at the screening visit.
* Best distance correction at screening in the range of spherical -1.50 D to +1.00 D inclusively and cylinder <= ±2.00 D with photopic high contrast binocular corrected distance visual acuity (CDVA) of 20/25 or better at the screening and baseline visits.
* Mesopic, high contrast binocular distance-corrected near visual acuity (DCNVA) no better than 20/40 (J3) at screening and baseline visits.

Exclusion Criteria:

- Presence of any ocular condition that, in the opinion of the investigator, could affect the safety of the participant or interpretation of efficacy parameters (e.g., uveitis, acute iritis, retinal detachment or retinal tear).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-09 (Estimated); Primary Completion 2023-04-04 (Estimated); Study Completion 2023-04-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 14 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (32):
- United States (32):
  - Trinity Research Group /ID# 243541, Dothan, Alabama
  - Arizona Eye Center /ID# 243897, Chandler, Arizona
  - Global Research Management /ID# 243544, Glendale, California
  - United Medical Research Institute /ID# 243531, Inglewood, California
  - Salvay Vision /ID# 243828, Newport Beach, California
  - The Eye Research Foundation /ID# 243524, Newport Beach, California
  - Sacramento Eye Consultants /ID# 243538, Sacramento, California
  - Nature Coast Clinical Research - Crystal River /ID# 243519, Crystal River, Florida
  - Segal Drug Trials, Inc /ID# 243521, Delray Beach, Florida
  - Eye Associates of Fort Meyers /ID# 243545, Fort Myers, Florida
  - Levenson Eye Associates Inc. /ID# 243532, Jacksonville, Florida
  - Emory University /ID# 243534, Atlanta, Georgia
  - Clayton Eye Clinical Research, LLC /ID# 243530, Morrow, Georgia
  - Coastal Research Associates /ID# 243525, Roswell, Georgia
  - Kannarr Eye Care /ID# 243542, Pittsburg, Kansas
  - Cincinnati Eye Institute- Edgewood /ID# 243810, Edgewood, Kentucky
  - The Eye Care Institute /ID# 243588, Louisville, Kentucky
  - Fraser Eye Center /ID# 244038, Fraser, Michigan
  - Silverstein Eye Centers /ID# 243546, Kansas City, Missouri
  - Eye Associates of North Jersey /ID# 243913, Dover, New Jersey
  - Northern New Jersey Eye Institute PA /ID# 243522, South Orange, New Jersey
  - Rochester Ophthalmological Group PC /ID# 243539, Rochester, New York
  - EyeCare Professionals Inc /ID# 243938, Powell, Ohio
  - Scott and Christie and Associates /ID# 243548, Cranberry Township, Pennsylvania
  - University Eye Surgeons /ID# 243926, Maryville, Tennessee
  - Advancing Vision Research /ID# 243529, Smyrna, Tennessee
  - Key-Whitman Eye Center /ID# 243928, Dallas, Texas
  - Eye associates /ID# 243526, San Antonio, Texas
  - Parkhurst Nuvision /ID# 244041, San Antonio, Texas
  - Hoopes, Durrie, Rivera Research /ID# 243535, Draper, Utah
  - Country Hills Eye Center /ID# 243520, Ogden, Utah
  - Southern Utah Medical Research /ID# 243931, St. George, Utah

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/